CLINICAL TRIAL: NCT04618458
Title: A Telehealth Diabetes Prevention Intervention for the Next Generation of African American Youth (TELE-GEN) Pilot Study
Brief Title: Telehealth Diabetes Prevention Intervention for African American Youth
Acronym: TELE-GEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Abigail Gamble, Assistant Professor, University of Mississippi Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AWD-000933; HHSN2682018000151 (Other Grant/Funding Number: Jackson Heart Study Community Engagement Center)
Record Dates: First submitted 2020-10-19; First posted 2020-11-06 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: PreDiabetes; Obesity; Obesity, Childhood
Keywords: prediabetic state; telehealth; healthy lifestyle; primary prevention; minority health
MeSH Terms: conditions — Prediabetic State; Obesity; Pediatric Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Eligible overweight/obese children and their overweight/obese parent (N=20 families) will receive the same telehealth diabetes prevention intervention based on Power to Prevent and delivered by a trained lifestyle coach. Families will meet weekly for 11-weeks (60-min sessions), and then monthly (60-min sessions) for 4 pilot behavioral reinforcement maintenance sessions (15 sessions total). Participants will meet in their respective groups (n=5 families per group) via videoconference using Wi-Fi-enabled tablets with cellular connectivity for the entire intervention. Sessions will consist of nutrition and physical activity behavior change strategies (20 min), problem solving and decision-making skills to circumvent barriers to behavioral change (20 min), and family goal setting and action planning (20 min). Assessment measures will be collected from the child and parent participants at baseline, 12-weeks (post-intervention), and 30-weeks (follow-up).
  Interventions: Behavioral: Power to Prevent

INTERVENTIONS:
Behavioral: Power to Prevent — Lifestyle diabetes prevention intervention based on the National Diabetes Prevention Program and tailored for African American families. The intervention will be delivered using telehealth and small group videoconferencing.

SUMMARY:
The Telehealth Diabetes Prevention Intervention for the Next Generation of African American Youth (TELE-GEN) pilot study will evaluate the implementation and early efficacy of a telehealth diabetes prevention intervention for African American (AA) children (8- to 11-years) and their parents. Power to Prevent is a lifestyle diabetes prevention intervention from the Centers for Disease Control and Prevention that is based on the Diabetes Prevention Program and tailored for AA families. To investigators knowledge, this intervention has not been evaluated in a clinical trial with AA families with children at risk for type 2 diabetes mellitus (T2DM), nor been delivered via telehealth. Employing an effectiveness-implementation hybrid study design, investigators aim to concurrently (1) conduct a single arm pilot trial to assess the early efficacy of Power to Prevent delivered via telehealth to treat overweight/obesity in AA children and their parent, while (2) evaluating an implementation strategy for the uptake of the intervention by the pediatric weight management clinic at the University of Mississippi Medical Center. The primary outcome will be stabilization or reduction in BMI z-score in children (index participant) and reduction in parent BMI (co-participant). Parents (n=20) will receive the same telehealth diabetes prevention intervention, which will be delivered by a racially concordant, trained Lifestyle Coach using small-group videoconferencing (5 parents per group). Sessions will consist of nutrition and physical activity behavior change strategies (20 min), problem solving and decision-making skills to circumvent barriers to behavioral change (20 min), and family goal setting and action planning (20 min). Child and parent measures will be assessed at baseline, 12-weeks (post-intervention), and 30-weeks (follow-up). The implementation strategy has two targets: (1) the pediatric weight management clinical and clinical care team; and (2) overweight/obese pediatric patients and their overweight/obese parents. The multifaceted implementation plan includes four discrete strategies: (1) creating a new clinical team; (2) changing the service site; (3) intervening with families; and (4) assessing organizational readiness. Preliminary findings will provide data to design a full-scale study that will include a powered pilot randomized controlled trial to test the interventions effectiveness for preventing T2DM, while evaluating a refined implementation protocol.

DETAILED DESCRIPTION:
The Telehealth Diabetes Prevention Intervention for the Next Generation of African American Youth (TELE-GEN) pilot study will evaluate the implementation and early efficacy of a telehealth diabetes prevention intervention for African American (AA) children (8- to 11-years-old) and their parents. Power to Prevent is a lifestyle diabetes prevention intervention from the Centers for Disease Control and Prevention that is based on the Diabetes Prevention Program (DPP) and tailored specifically for AA families. To the knowledge of the study's investigators, this intervention has not yet been evaluated in a clinical trial with AA families with children at risk for T2DM, nor been delivered via telehealth. Employing an effectiveness-implementation hybrid research design, investigators aim to concurrently: (1) conduct a single arm pilot clinical trial to assess the early efficacy of Power to Prevent delivered via telehealth to treat overweight/obesity in AA children and their parent, while (2) comprehensively evaluate a multifaceted implementation strategy for the uptake of Power to Prevent delivered via telehealth by UMMC's pediatric weight management clinic. The primary outcome measure will be stabilization or reduction in BMI z-score in children (index participant) and a reduction in parent BMI (co-participant). Eligible overweight/obese children and their overweight/obese parent (N=20 families) will receive the same telehealth diabetes prevention intervention based on Power to Prevent, which will be delivered by a racially concordant Lifestyle Coach trained in the DPP. Families will meet weekly for 11-weeks (60-min sessions), and then monthly (60-min sessions) for 4 pilot behavioral reinforcement maintenance sessions (15 sessions total). Participants will meet in their respective groups (n=5 families per group) via videoconferencing using Wi-Fi-enabled tablets with cellular connectivity for the entire intervention. Sessions will consist of nutrition and physical activity behavior change strategies (20 min), problem solving and decision-making skills to circumvent barriers to behavioral change (20 min), and family goal setting and action planning (20 min). Assessment measures will be collected from the child and parent participants at baseline, 12-weeks (post-intervention), and 30-weeks (follow-up). The implementation strategy has two targets: (1) UMMC's pediatric weight management clinical setting and clinical care team; and (2) overweight/obese pediatric patients and their overweight/obese parents referred to and engaged in intensive obesity treatment for the prevention of T2DM. The multifaceted implementation plan includes four discrete strategies: (1) creating a new clinical team; (2) changing the service site; (3) intervening with families; and (4) assessing organizational readiness. Preliminary findings will provide sufficient data to design a full-scale effectiveness-implementation hybrid study that will include a powered pilot randomized controlled trial (RCT) to test the interventions effectiveness for preventing T2DM, while evaluating a refined implementation protocol. The overall purpose of the TELE-GEN pilot study directly contributes to the goal of the Jackson Heart Study Community Engagement Center by leveraging existing infrastructure and technology to engage AA families in a virtual community to prevent T2DM. The proposed aims and methods also parallel the NHLBI's strategic goal to advance transnational research.

ELIGIBILITY:
Inclusion Criteria:

* AA parents (biological, grandparent, legal guardian) and their 8- to 11-year-old child residing in the same home.
* One overweight/obese parent (BMI ≥25 kg/m2) and child (≥ 85th% age-/sex-specific BMI).
* Parent at-risk for diabetes (American Diabetes Association risk test) AND HbA1c 5.7% - 6.4%.

Exclusion Criteria:

* child or parent has a history of T2DM or a screening HbA1c >6.4%;
* is taking glucose-lowering medications;
* is participating in a supervised weight loss program;
* is pregnant or breast feeding;
* has conditions limiting participation;
* has undergone weight loss surgery;
* is moving out-of-state within 6 months.
* If a parent becomes pregnant during the study, we will include only child data (index participant) in analyses

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-18 (Actual)

PRIMARY OUTCOMES:
Child BMI z-score | Change from baseline child BMI z-score to 12-weeks
  Standard anthropometric procedures and a calibrated body weight scale (Seca 777 digital scale with stadiometer) will be used to measure participants' weight (0.1kg), stature (0.1 cm); child BMI percentile will be calculated using the statistic equations made available on the Centers for Disease Control and Prevention (CDC) website
Child BMI z-score | Change from baseline child BMI z-score to 30-weeks
  Standard anthropometric procedures and a calibrated body weight scale (Seca 777 digital scale with stadiometer) will be used to measure participants' weight (0.1kg), stature (0.1 cm); child BMI percentile will be calculated using the statistic equations made available on the CDC website
Parent BMI | Change from baseline parent BMI to 12-weeks
  Standard anthropometric procedures and a calibrated body weight scale will be used to measure participants' weight (0.1kg), stature (0.1 cm); after converting cm to m, BMI = kg/m2
Parent BMI | Change from baseline parent BMI to 30-weeks
  Standard anthropometric procedures and a calibrated body weight scale will be used to measure participants' weight (0.1kg), stature (0.1 cm); after converting cm to m, BMI = kg/m2

SECONDARY OUTCOMES:
Child physical activity | Change from baseline child physical activity to 12-weeks
  Objective assessment using ActiGraph GT9X Link Accelerometers; child and parent will wear accelerometer continuously for seven day period
Child physical activity | Change from baseline child physical activity to 30-weeks
  Objective assessment using ActiGraph GT9X Link Accelerometers; child and parent will wear accelerometer continuously for seven day period
Parent physical activity | Change from baseline parent physical activity to 12-weeks
  Objective assessment using ActiGraph GT9X Link Accelerometers; child and parent will wear accelerometer continuously for seven day period
Parent physical activity | Change from baseline parent physical activity to 30-weeks
  Objective assessment using ActiGraph GT9X Link Accelerometers; child and parent will wear accelerometer continuously for seven day period
Child out-of-school sedentary time | Change from baseline in child out-of-school sedentary time to 12-weeks
  Objective assessment using ActiGraph GT9X Link Accelerometers; child and parent will wear accelerometer continuously for seven day period
Child out-of-school sedentary time | Change from baseline in child out-of-school sedentary time to 30-weeks
  Objective assessment using ActiGraph GT9X Link Accelerometers; child and parent will wear accelerometer continuously for seven day period
Parent sedentary time | Change from baseline in parent sedentary time to 12-weeks
  Objective assessment using ActiGraph GT9X Link Accelerometers; child and parent will wear accelerometer continuously for seven day period
Parent sedentary time | Change from baseline in parent sedentary time to 30-weeks
  Objective assessment using ActiGraph GT9X Link Accelerometers; child and parent will wear accelerometer continuously for seven day period
Child Hemoglobin A1c | Change from baseline child Hemoglobin A1c to 12-weeks
  A1CNOW+ System for reliable point-of-care HbA1c measurement; non-fasting 5 μL blood
Child Hemoglobin A1c | Change from baseline child Hemoglobin A1c to 30-weeks
  A1CNOW+ System for reliable point-of-care HbA1c measurement; non-fasting 5 μL blood
Parent Hemoglobin A1c | Change from baseline parent Hemoglobin A1c to 12-weeks
  A1CNOW+ System for reliable point-of-care HbA1c measurement; non-fasting 5 μL blood
Parent Hemoglobin A1c | Change from baseline parent Hemoglobin A1c to 30-weeks
  A1CNOW+ System for reliable point-of-care HbA1c measurement; non-fasting 5 μL blood
Child systolic blood pressure | Change from baseline child systolic blood pressure to 12-weeks
  Welch Allyn blood pressure unit following the American Heart Association guidelines for children.
Child diastolic blood pressure | Change from baseline child diastolic blood pressure to 12-weeks
  Welch Allyn blood pressure unit following the American Heart Association guidelines for children.
Child systolic blood pressure | Change from baseline child systolic blood pressure to 30-weeks
  Welch Allyn blood pressure unit following the American Heart Association guidelines for children.
Child diastolic blood pressure | Change from baseline child diastolic blood pressure to 30-weeks
  Welch Allyn blood pressure unit following the American Heart Association guidelines for children.
Parent systolic blood pressure | Change from baseline parent systolic blood pressure to 12-weeks
  Welch Allyn blood pressure unit following the American Heart Association guidelines for adults.
Parent diastolic blood pressure | Change from baseline parent diastolic blood pressure to 12-weeks
  Welch Allyn blood pressure unit following the American Heart Association guidelines for adults.
Parent systolic blood pressure | Change from baseline in parent systolic blood pressure to 30-weeks
  Welch Allyn blood pressure unit following the American Heart Association guidelines for adults.
Parent diastolic blood pressure | Change from baseline in parent diastolic blood pressure to 30-weeks
  Welch Allyn blood pressure unit following the American Heart Association guidelines for adults.
Child resting heart rate | Change from baseline in child resting heart rate to 12-weeks
  Welch Allyn blood pressure unit
Child resting heart rate | Change from baseline in child resting heart rate to 30-weeks
  Welch Allyn blood pressure unit
Parent resting heart rate | Change from baseline in parent resting heart rate to 12-weeks
  Welch Allyn blood pressure unit
Parent resting heart rate | Change from baseline in parent resting heart rate to 30-weeks
  Welch Allyn blood pressure unit
Parent readiness to change | Change from baseline in parent readiness to change to 12-weeks
  Adapted from Rhee et al., a 6-item instrument to assess parents readiness and intentions to make dietary, physical activity and sedentary changes.
Parent readiness to change | Change from baseline in parent readiness to change to 30-weeks
  Adapted from Rhee et al., a 6-item instrument to assess parents readiness and intentions to make dietary, physical activity and sedentary changes.
Parent self-efficacy | Change from baseline in parent self-efficacy to 12-weeks
  Valid and reliable (Norma et al., 2018) 14-item instrument to measure parent efficacy for influencing children's physical activity, sedentary behavior and dietary behavior using an 11-point Likert scale; 0-not confident, 10-absolutely confident.
Parent self-efficacy | Change from baseline in parent self-efficacy to 30-weeks
  Valid and reliable (Norma et al., 2018) 14-item instrument to measure parent efficacy for influencing children's physical activity, sedentary behavior and dietary behavior using an 11-point Likert scale; 0-not confident, 10-absolutely confident.
Child self-efficacy | Change from baseline in child self-efficacy to 12-weeks
  A 9-item valid and reliable instrument by Lassetter et al., 2014 asking children to report their confidence on a 3-point Likert scale for eating healthy and being physically active; 1 item added to assess efficacy for watching less than 2 hours of television (TV) every day.
Child self-efficacy | Change from baseline in child self-efficacy to 30-weeks
  A 9-item valid and reliable instrument by Lassetter et al., 2014 asking children to report their confidence on a 3-point Likert scale for eating healthy and being physically active; 1 item added to assess efficacy for watching less than 2 hours of TV every day.
Parent perceived family functioning | Change from baseline in parent perceived family functioning to 12-weeks
  McMaster Family Assessment Device; a valid and reliable 60-item instrument using a 4-point Likert scale; subscales include problem solving, communication, roles, affective responsiveness, affective involvement, behavior control, general functioning
Parent perceived family functioning | Change from baseline in parent perceived family functioning to 30-weeks
  McMaster Family Assessment Device; a valid and reliable 60-item instrument using a 4-point Likert scale; subscales include problem solving, communication, roles, affective responsiveness, affective involvement, behavior control, general functioning
Home physical activity and food environment | Change from baseline in parent perceived home physical activity and food environment to 12-weeks
  The Home Environment Survey; valid and reliable instrument (Gattshall et al., 2008) to measure the physical and social environment for food and physical activity; modified to include the physical and social environment for TV time (sedentary behavior); modified to include 79-items total; Dimensions: physical activity availability and accessibility of physical activity equipment, technology and food (i.e. fruit and vegetables); parental role modeling of physical activity, sedentary behavior, and dietary behavior.
Home physical activity and food environment | Change from baseline in parent perceived home physical activity and food environment to 30-weeks
  The Home Environment Survey; valid and reliable instrument (Gattshall et al., 2008) to measure the physical and social environment for food and physical activity; modified to include the physical and social environment for TV time (sedentary behavior); modified to include 79-items total; Dimensions: physical activity availability and accessibility of physical activity equipment, technology and food (i.e. fruit and vegetables); parental role modeling of physical activity, sedentary behavior, and dietary behavior.
Parent perceived child obesity-related behavior | Change from baseline in parent perceived child health behavior to 12-weeks
  Child Obesity Behavior Scale; adapted from Rhee et al., 2014; 20-items to measure food, physical activity and sedentary behavior quantity and frequency.
Parent perceived child obesity-related behavior | Change from baseline in parent perceived child health behavior to 30-weeks
  Child Obesity Behavior Scale; adapted from Rhee et al., 2014; 20-items to measure food, physical activity and sedentary behavior quantity and frequency.
Child perceived obesity-related behavior | Change from baseline in child health behavior to 12-weeks
  Healthy Eating and Physical Activity Recall Questionnaire; 9-items (Lassettter et al., 2017); modified to include questions for sedentary environment; 5-items.
Child perceived obesity-related behavior | Change from baseline in child health behavior to 30-weeks
  Healthy Eating and Physical Activity Recall Questionnaire; 9-items (Lassettter et al., 2017); modified to include questions for sedentary environment; 5-items.
Neighborhood Perception Survey | Change from baseline in parent neighborhood perception to 12-weeks
  Valid and reliable 31-item instrument used by Mujahod et al., 2007 to assess 7 dimensions of neighborhood: aesthetic quality, walking environment, availability of healthy foods, safety, violence, social cohesion, activities with neighbors.
Neighborhood Perception Survey | Change from baseline in parent neighborhood perception to 30-weeks
  Valid and reliable 31-item instrument used by Mujahod et al., 2007 to assess 7 dimensions of neighborhood: aesthetic quality, walking environment, availability of healthy foods, safety, violence, social cohesion, activities with neighbors.
Child waist circumference | Change from baseline in child waist circumference to 12-weeks
  A Seca 203 circumference measuring tape will be used to assess participants waist circumference.
Child waist circumference | Change from baseline in child and parent waist circumference to 30-weeks
  A Seca 203 circumference measuring tape will be used to assess participants waist circumference.
Parent waist circumference | Change from baseline in parent waist circumference to 12-weeks
  A Seca 203 circumference measuring tape will be used to assess participants waist circumference.
Parent waist circumference | Change from baseline in parent waist circumference to 30-weeks
  A Seca 203 circumference measuring tape will be used to assess participants waist circumference.
Parent stress | Change from baseline in parent stress to 12-weeks
  Perceived Stress Scale; 10-items (Cohen, 1994)
Parent stress | Change from baseline in parent stress to 30-weeks
  Perceived Stress Scale; 10-items (Cohen, 1994)
Child stress | Change from baseline in parent stress to 12-weeks
  PROMIS Pediatric Psychological and Physical Stress Scale; 19-items and 26-items (Bevans et al., 2018)
Child stress | Change from baseline in parent stress to 30-weeks
  PROMIS Pediatric Psychological and Physical Stress Scale; 19-items and 26-items (Bevans et al., 2018)

OTHER OUTCOMES:
Child tanner stage | Change from baseline in child tanner stage to 12-weeks
  A valid and reliable self-administered rating scale for pubertal development; 5-items. (Carskadon and Acebo, 1993)
Child tanner stage | Change from baseline in child tanner stage to 30-weeks
  A valid and reliable self-administered rating scale for pubertal development; 5-items. (Carskadon and Acebo, 1993)

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Gamble, PhD, MS, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gamble A, Beech BM, Wade BC, Sutton VD, Lim C, Sandridge S, Welsch MA. Telehealth Diabetes Prevention Intervention for the Next Generation of African American Youth: Protocol for a Pilot Trial. JMIR Res Protoc. 2021 Mar 31;10(3):e25699. doi: 10.2196/25699. PMID 33787504
- See also: TELE-GEN Protocol — https://www.researchprotocols.org/2021/3/e25699